CLINICAL TRIAL: NCT04475679
Title: Clinical Evaluation of a New Dual Cure Universal Adhesive (Adhese Universal DC) in the Indirect Restorative Therapy: A Randomised, Controlled Clinical Trial
Brief Title: Clinical Evaluation of Adhese Universal DC in the Indirect Restorative Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not sufficient cases for recall to investigate performance of test product
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LL3615088
Record Dates: First submitted 2020-07-08; First posted 2020-07-17 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Dental Caries; Defective Tooth Restorations
Keywords: caries; restoration
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adhese Universal DC (Experimental)
  Interventions: Device: Adhese Universal DC
- Adhese Universal (Active Comparator)
  Interventions: Device: Adhese Universal

INTERVENTIONS:
Device: Adhese Universal DC — Adhese Universal DC, a dental adhesive, will be used in conjunction with the luting cement Variolink Esthetic DC to bond indirect restorations to the tooth surface
  Arms: Adhese Universal DC
Device: Adhese Universal — Adhese Universal, a dental adhesive, will be used in conjunction with the luting cement Variolink Esthetic DC to bond indirect restorations to the tooth
  Arms: Adhese Universal

SUMMARY:
A post market clinical follow up study (PMCF) with Adhese Universal DC is planned to ensure the safety and efficacy of the product. It is a study with two arms. Inlays and onlays for molars and premolars will be luted with Adhese Universal DC or Adhese Universal.

DETAILED DESCRIPTION:
This study aims to assess the long-term safety of Adhese Universal DC in terms of tooth vitality and failure rate of placed restorations. Tooth vitality is an indicator for the health status of the dental pulp. A vitality test is performed to acquire information about the vitality of teeth. A healthy dental pulp offers a positive response to the vitality test. Once the dental pulp is injured an irreversible inflammatory reaction starts with a possible necrosis of the dental pulp. Pulpa necrosis is followed by a negative response to the vitality test.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Indication for indirect restorations (inlay, onlay) in molar or premolar - replacement of insufficient fillings (e.g. due to caries at margins, filling fracture, fracture of the tooth, poor quality of the surface, leaking margin, etc.) or extensive primary caries
* The occlusal area of the restoration must cover at least 1/3 of the occlusal area of the tooth.
* Participant wishes a restoration within the scope of the study (signed informed consent after detailed explanation and study of the patient information)
* 2-operative discomfort of the tooth to be restored should not exceed 3 on the visual analogue scale (VAS) (0=no pain, 10=maximum conceivable pain) due to temperature stimulus or bite sensitivity
* Max. 2 restorations per participant in different quadrants.
* Vital tooth
* Healthy periodontium, no active periodontitis
* Contact with adjacent teeth (at least at one side) and opposing teeth present with at least one contact point.
* Sufficient language skills

Exclusion Criteria:

* Sufficient isolation not possible, dry working field cannot be guaranteed
* Participants with a proven allergy to one of the ingredients of the materials used
* Participants with proven allergy to local anaesthetics
* High caries activity/ poor oral hygiene
* Participants with severe systemic diseases
* Pregnancy
* Nonvital tooth or tooth with irreversible pulpitis
* Indication for direct pulp capping
* Symptoms of SARS-CoV2 infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ivoclar Vivadent, Schaan, Liechtenstein

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period took place between 14.09.2020-30.06.2021 in the clinic.
Groups:
- Adhese Universal DC: Adhese Universal DC: Adhese Universal DC, a dental adhesive, will be used in conjunction with the luting cement Variolink Esthetic to bond indirect restorations to the tooth surface
- Adhese Universal: Adhese Universal: Adhese Universal, a dental adhesive, will be used in conjunction with the luting cement Variolink Esthetic to bond indirect restorations to the tooth
Period: Overall Study
Arm/Group | Adhese Universal DC | Adhese Universal
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adhese Universal DC | Adhese Universal | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Customized [Count of Participants; unit: Participants]
  18-65 years | 40 | 40 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 27 | 25 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: FDI 11 Postoperative Hypersensitivity After Inlay/Onlay Restoration, FDI Score 1-5
Description: assessed by tests with thermal stimuli and occlusal forces (during biting) determined by VAS (Visual Analog Scale) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: Baseline (7-10 days)
Population: Baseline
Measure: Number; unit: Inlays/Onlays
Units Other Than Participants: Inlays/Onlays
Arm/Group | Adhese Universal DC | Adhese Universal
Number analyzed (Participants) | 39 | 39
Number analyzed (Inlays/Onlays) | 39 | 39
Inlays/Onlays
  FDI 11 (Postoperative hypersensitivity), FDI Score 1 | 39 | 38
  FDI 11 (Postoperative hypersensitivity), FDI Score 2 | 0 | 1
  FDI 11 (Postoperative hypersensitivity), FDI Score 3-5 | 0 | 0

2. Primary Outcome: FDI 11 Postoperative Hypersensitivity After Inlay/Onlay Restorations, FDI Score 1-5
Description: as for outcome 1
Time Frame: 12 months
Population: Baseline
Measure: Number; unit: Inlays/Onlays
Units Other Than Participants: Inlays/Onlays
Arm/Group | Adhese Universal DC | Adhese Universal
Number analyzed (Participants) | 37 | 36
Number analyzed (Inlays/Onlays) | 37 | 36
Inlays/Onlays
  FDI 11 (Postoperative hypersensitivity), FDI Score 1 | 37 | 36
  FDI 11 (Postoperative hypersensitivity), FDI Score 2 | 0 | 0
  FDI 11 (Postoperative hypersensitivity), FDI Score 3-5 | 0 | 0

3. Secondary Outcome: Vitality of Restored Teeth After Inlay/Onlay Restorations, FDI Score 1-5
Description: assessed by a cold stimuli test on the patient teeth (cotton pellet and refrigerating spray) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: Baseline
Measure: Number; unit: restored teeth
Units Other Than Participants: restored teeth
Arm/Group | Adhese Universal DC | Adhese Universal
Number analyzed (Participants) | 40 | 40
Number analyzed (restored teeth) | 40 | 40
restored teeth
  Vitality, FDI Score 1 | 40 | 40
  Vitality, FDI Score 2-5 | 0 | 0

4. Secondary Outcome: FDI 13 Fracture of Restored Teeth After Inlay/Onlay Restorations, FDI Score 1-5
Description: assessed on patient teeth by checking tooth integrity (looking for enamel cracks, tooth fractures) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: Baseline
Measure: Number; unit: restored Teeth
Units Other Than Participants: restored Teeth
Arm/Group | Adhese Universal DC | Adhese Universal
Number analyzed (Participants) | 40 | 40
Number analyzed (restored Teeth) | 40 | 40
restored Teeth
  FDI 13 (Tooth Integrity), FDI Score 1 | 40 | 40
  FDI 13 (Tooth Integrity), FDI Score 2-5 | 0 | 0

5. Secondary Outcome: FDI 5 Retention/Fracture of Restorations After Inlays/Onlays Restorations, FDI Score 1-5
Description: assessed on patient teeth (checking inlays/onlays for fractures, cracks, small hairline cracks, chip fractures, material damage) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: Baseline
Measure: Number; unit: Inlays/Onlays
Units Other Than Participants: Inlays/Onlays
Arm/Group | Adhese Universal DC | Adhese Universal
Number analyzed (Participants) | 40 | 40
Number analyzed (Inlays/Onlays) | 40 | 40
Inlays/Onlays
  Fracture of material and retention, FDI Score 1 | 39 | 38
  Fracture of material and retention, FDI Score 2 | 0 | 0
  Fracture of material and retention, FDI Score 3 | 0 | 1
  Fracture of material and retention, FDI Score 4 | 0 | 0
  Fracture of material and retention, FDI Score 5 | 1 | 1

6. Secondary Outcome: FDI 6 Marginal Quality After Inlay/Onlay Restorations, FDI Score 1-5
Description: assessed on the patient teeth (looking for marginal gaps/Fractures, checking outlines) following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable"
Time Frame: Baseline
Measure: Number; unit: Inlays/Onlays
Units Other Than Participants: Inlays/Onlays
Arm/Group | Adhese Universal DC | Adhese Universal
Number analyzed (Participants) | 39 | 39
Number analyzed (Inlays/Onlays) | 39 | 39
Inlays/Onlays
  Marginal Quality, FDI Score 1 | 37 | 37
  Marginal Quality, FDI Score 2 | 2 | 2
  Marginal Quality, FDI Score 3-5 | 0 | 0

7. Secondary Outcome: Vitality of Restored Teeth After Inlay/Onlay Restorations, FDI Score 1-5
Description: as for outcome 3
Time Frame: 12 months
Measure: Number; unit: restored teeth
Units Other Than Participants: restored teeth
Arm/Group | Adhese Universal DC | Adhese Universal
Number analyzed (Participants) | 40 | 40
Number analyzed (restored teeth) | 40 | 40
restored teeth
  Vitality, FDI Score 1 | 40 | 40
  Vitality, FDI Score 2-5 | 0 | 0

8. Secondary Outcome: FDI 13 Fracture of Restored Teeth After Inlay/Onlay Restorations, FDI Score 1-5
Description: as for outcome 4
Time Frame: 12 months
Measure: Number; unit: restored teeth
Units Other Than Participants: restored teeth
Arm/Group | Adhese Universal DC | Adhese Universal
Number analyzed (Participants) | 40 | 40
Number analyzed (restored teeth) | 40 | 40
restored teeth
  FDI 13 (Tooth Integrity), FDI Score 1 | 40 | 40
  FDI 13 (Tooth Integrity), FDI Score 2-5 | 0 | 0

9. Secondary Outcome: FDI 5 Retention/Fracture of Restorations After Inlays/Onlays Restorations, FDI Score 1-5
Description: as for outcome 5
Time Frame: 12 months
Measure: Number; unit: Inlays/Onlays
Units Other Than Participants: Inlays/Onlays
Arm/Group | Adhese Universal DC | Adhese Universal
Number analyzed (Participants) | 40 | 40
Number analyzed (Inlays/Onlays) | 40 | 40
Inlays/Onlays
  Fracture of material and retention,FDI Score 1 | 37 | 36
  Fracture of material and retention,FDI Score 2-4 | 0 | 0
  Fracture of material and retention,FDI Score 5 | 3 | 4

10. Secondary Outcome: FDI 6 Marginal Quality After Inlay/Onlay Restorations, FDI Score 1-5
Description: as for outcome 6
Time Frame: 12 months
Measure: Number; unit: Inlays/Onlays
Units Other Than Participants: Inlays/Onlays
Arm/Group | Adhese Universal DC | Adhese Universal
Number analyzed (Participants) | 37 | 36
Number analyzed (Inlays/Onlays) | 37 | 36
Inlays/Onlays
  Marginal Quality, FDI Score 1 | 37 | 36
  Marginal Quality, FDI Score 2-5 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: An adverse event was defined as something unfavourable that happened to the treated tooth and was reported as part of the regular recall by the investigator.
  (either technical AE such as fracture of the treated tooth or restoration/tooth replacement and retention loss of the restoration/tooth replacement, or biological AE such as post-operative sensitivity and secondary caries on the treated tooth)
Arm/Group | Adhese Universal DC | Adhese Universal
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 3/40 | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adhese Universal DC (N=40) | Adhese Universal (N=40)
Retention Loss (Product Issues) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT04475679/Prot_SAP_000.pdf